CLINICAL TRIAL: NCT01629212
Title: Comparative and Analytical Study for Effectiveness and Safety of Tiropramide HCl and Octylonium Bromide in the Treatment of Irritable Bowel Syndrome: Mullticenter, Randomized, Double Blind, Active Controlled Study
Brief Title: Comparison of the Efficacy and Safety of Tiropramide and Octylonium in the Treatment of Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: DW-TRP001
Record Dates: First submitted 2012-06-21; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — octylonium

ARMS (2):
- Tiropramide HCl (Experimental)
  Interventions: Drug: Tiropramide HCl 100mg
- Octylonium bromide (Active Comparator)
  Interventions: Drug: Octylonium bromide 20mg

INTERVENTIONS:
Drug: Tiropramide HCl 100mg
  Arms: Tiropramide HCl
Drug: Octylonium bromide 20mg
  Arms: Octylonium bromide

SUMMARY:
The purpose of this study was to compare the Efficacy and Safety of Tiropramide HCl and Octylonium bromide in the Treatment of Irritable Bowel Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 20-75 years)
2. Patients who had been suffered from IBS as defined by Rome III criteria
3. Patients who had abdominal pain at least 2 days/week, during the run-in period of 2 weeks

Exclusion Criteria:

1. Patients with known intolerance to tiropramide or octylonium
2. Patients with uncontrolled diabetes, uncontrolled hypertension or thyroid dysfunction
3. Patients who had the history of cancer [However, patients with cancer other than gastrointerstinal cancer, who have not recurr within 5 years after treatment were possible for enrollment]
4. Patients with hepatic or renal dysfunction
5. Patients with lactose intorelance

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2011-12; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Change of abdominal pain VAS scores from baseline to week 4

SECONDARY OUTCOMES:
Change of abdominal pain VAS scores from baseline to week 2
Change of abdominal discomfort VAS scores from baseline to week 2 and 4

CONTACTS AND LOCATIONS:
Locations (1):
- Han Yang University Hospital, Seoul, South Korea